CLINICAL TRIAL: NCT02227953
Title: A Pilot Study for the Improvement of Cognitive Function (ADAS-Cog 11) After Transcranial Direct Current Stimulation in Mild to Moderate Alzheimer's Disease
Brief Title: A Pilot Study of tDCS for Mild to Moderate Alzhemier's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Collaborators: Ybrain Inc. (Industry)
Responsible Party: Principal Investigator, Duk Lyul Na, Professor of Neurology, Sungkyunkwan University School of Medicine, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SMC 2014-04-025
Record Dates: First submitted 2014-08-26; First posted 2014-08-28 (Estimated); Last update posted 2014-09-03 (Estimated); Status verified 2014-08

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's Disease; AD; tDCS; transcranial direct current stimulation
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- YBand (YDT-201N) (Experimental): transcranial Direct Current Stimulation (tDCS) application 7 days a week for 12 weeks (total of 84 applications)
  Interventions: Device: Yband (YDT-201N)
- sham-Yband (YDT-201N) (Sham Comparator): sham-tDCS application 7 days a week for 12 weeks (total of 84 applications)
  Interventions: Device: sham-Yband (YDT-201N)

INTERVENTIONS:
Device: Yband (YDT-201N) — transcranial Direct Current Stimulation (tDCS) 2mA for 30 min; 20 sec of ramp-up and -down; left (anode) and right (cathode) Dorsolateral prefrontal cortex (DLPFC)
  Arms: YBand (YDT-201N)
Device: sham-Yband (YDT-201N) — transcranial Direct Current Stimulation (tDCS) 2mA for 20 sec; left (anode) and right (cathode) Dorsolateral prefrontal cortex (DLPFC)
  Arms: sham-Yband (YDT-201N)

SUMMARY:
The primary objective of this preliminary study is to investigate whether the transcranial direct current stimulation (tDCS) improves the cognitive function in patients with Alzheimer's disease

DETAILED DESCRIPTION:
Twenty patients were recruited and randomized to receive either real or sham-tDCS over the left (anode) and right (cathode) dorsolateral prefrontal cortex (DLPFC). Their legally responsible caregivers were provided with mobile tDCS device, and were instructed to use it on the patients at home. 30-minute session of the stimulation were applied everyday in the morning for 12 weeks. The patients were evaluated at baseline, at week 6 and 12.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have Korean version of Mini Mental Status Examination score 10 to 24
* Subjects who have SVLT and RCFT delayed recall test scores lower than 1.5SD
* Subjects who have had other cognitive impairments besides memory
* Subjects who have Seoul-Instrumental Activities of Daily Living score (S-IADL) of 8 or more.
* Subjects who are only dementia of Alzheimer's type
* Subjects who are right-handed
* Subjects who are able to read and write
* Both patient and legally responsible caregiver has provided informed consent
* According to the latest MRI result, periventricular white matter cap or band is less than 10mm, or the deep white matter hyper-intensity is less than 25 mm

Exclusion Criteria:

* Subjects who have a history of stroke and seizures
* Subjects who have any illnesses that may disturb the patients completing the trials, including stroke, Parkinson's disease, type 1 diabetes, uncontrollable high blood pressure, Huntington's disease, cerebral palsy, liver failure, nephritis, encephalitis, meningitis, scleroma, seizures and a transient ischemic attack.
* Subjects who have a History of DSM-IV Axis I disorders
* Subjects who have neurologic problems on physical examination that cause memory disturbances
* Subjects who have Extremely sensitive skin
* Subjects who have suffered from the cancer in 3 years
* Subjects who have had a cerebrovascular neurosurgery in medical history
* Subjects who have dyspnea in sitting position
* Subjects who have problems with memory, language and problem-solving for 2 hours after the heart attack.
* Subjects who have a history of drug or alcohol abuse (in the past 5 years)
* Subjects who have a history of mental or emotional disorders (in the past 5 years)
* Subjects who have been lapsed into unconsciousness for an hour because of other reasons than general anesthesia
* Subjects who have a history of hospitalization due to head injury
* Subjects who are unable to read even with glasses
* Subjects who are unable to understand the conversation due to the hearing defect (even with the hearing aid)

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-08; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Change in cognitive function | from baseline to Week 6 and Week 12
  Measured by ADAS-Cog 11

SECONDARY OUTCOMES:
Change in questionnaire | from baseline to Week 12
  Measured by I-PAQ (International Physical Activity Questionnaire), Quality of Life Scale, KDSQ (Korean Dementia Screening Questionnaire), and Prospective and retrospective memory questionnaire
Change in cognitive function | from baseline to Week 6 and Week 12
  Measured by Korean version of Montreal Cognitive Assessment (K-MoCA), Korean version of Mini Mental Status Examination (K-MMSE), and Clinical Dementia Rating - Sum of Boxes(CDR-SOB)
Change in Korean version of Geriatric Depression Scale (K-GDS) | from baseline to Week 6 and Week 12
Change in activities of daily living | from baseline to Week 12
  Measured by Korean version of Bayer ADL (K-ADL) and S-IADL (Seoul-Instrumental Activities of Daily Living score)
Change in behavioral symptoms | from baseline to Week 6 and Week 12
  Measured by Neuropsychiatric Inventory
Change in Clinician's Interview-Based Impression of Change Plus (CIBIC plus) | from baseline to Week 12
Change in tDCS feedback | Week 2, 4, 6 and 12
  Measured by tDCS feedback questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Duk L. Na, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea